CLINICAL TRIAL: NCT03731442
Title: Salvage Chemoradiation Therapy for Recurrence After Radical Surgery or Palliative Surgery in Esophageal Cancer Patients: A Prospective, Multicenter Clinical Trial
Brief Title: Salvage Chemoradiation Therapy for Recurrence After Radical Surgery or Palliative Surgery in Esophageal Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Anyang Tumor Hospital (Other); Fujian Cancer Hospital (Other Government); Peking University Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-175/1753
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Cancer
Keywords: Salvage therapy; Recurrence; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms; Recurrence | interventions — Paclitaxel; Platinum; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involved field irradiation (Experimental): Patients after R0 surgery whose recurrence lesion larger than 5cm in diameter, or largest diameter was less than 5cm but with skip metastasis far from primary tumor or their time-to-recurrence longer than 16 months were assigned to involved field irradiation group. For lesions far from the thoracic stomach, the prescribed dose is 60Gy/2Gy/30f, and for lesions close to the thoracic stomach, the prescribed dose is 59.4-61.2Gy/1.8Gy/33-34f. Chest CT scan is planned at 50Gy. Radiation field should be modified according to the tumor response. Concurrent chemotherapy of paclitaxel and platinum was delivered every 3 weeks. PEG-rhG-CSF (3-6mg) should be given after 48 hours of chemotherapy.If patients received postoperative chemotherapy of paclitaxel and platinum and went through local-regional recurrence within six months, it is allowed to deliver chemotherapy regimens in the second line. Consolidate chemotherapy were adjusted to the patients after radiation therapy.
  Interventions: Radiation: Involved field irradiation; Drug: Paclitaxel; Drug: Platinum; Drug: PEG-rhG-CSF
- Elective field irradiation (Experimental): Patients after R1/R2 surgery or R0 surgery with the recurrence lesion whose diameter was less than 5cm without skip metastasis far from primary tumor and time-to-recurrence shorter than 16 months were assigned to elective field irradiation group. For lesions far from the thoracic stomach, the prescribed dose is 50.4Gy/1.8Gy/28f with a simultaneously integrated boost up to 59.92-62.16Gy/2.14-2.22Gy/28f. For lesions close to the thoracic stomach, the prescribed dose is 50.4Gy/1.8Gy/28f with a sequential boost of 10-12Gy/1.8-2Gy/5-7f. For patients whose planned thoracic stomach V50>50%, the dose should be lowered to 45Gy/1.8Gy/25f. Concurrent chemotherapy of paclitaxel and platinum was delivered every 3 weeks. PEG-rhG-CSF should be given in need. If patients received postoperative chemotherapy of TP and went through local-regional recurrence within 6 months, chemotherapy regimens delivered in the second line. Consolidate chemotherapy were adjusted to the patients after radiation therapy.
  Interventions: Radiation: Elective field irradiation; Drug: Paclitaxel; Drug: Platinum; Drug: PEG-rhG-CSF

INTERVENTIONS:
Radiation: Involved field irradiation — Involved field irradiation; intensity-modulated radiation therapy
  Arms: Involved field irradiation
Radiation: Elective field irradiation — Elective field irradiation; intensity-modulated radiation therapy
  Arms: Elective field irradiation
Drug: Paclitaxel — Paclitaxel 135-150mg/m2, d1, every 3 weeks
Drug: Platinum — for lobaplatin, 30mg/m2, d1-2, total dose should not exceed 50mg,every 3 weeks; for nedaplatin 50mg/m2, d1-2, every 3 weeks;
Drug: PEG-rhG-CSF — PEG-rhG-CSF 3-6mg, 48 hours after chemotherapy

SUMMARY:
Currently, adjuvant therapy is not recommended for patients with esophageal squamous cell carcinoma who received radical surgery. However, the recurrence rate is as high as 23.8%-58%, and the median time-to-recurrence is about 10.5 months. In patients who had residual tumor after surgery, evidence lacks for chemoradiation. The aim of the study is to evaluate the efficacy and safety of chemoradiation therapy in patients with recurrences after radical surgery or palliative surgery.

DETAILED DESCRIPTION:
Currently, adjuvant therapy is not recommended for patients with esophageal squamous cell carcinoma who received surgery as their first treatment. However, the recurrence rate is as high as 23.8%-58%, and the median time-to-recurrence is about 10.5 months. In patients who had residual tumor after surgery, evidence lacks for chemoradiation.

Retrospective data of 218 cases in our hospital indicated patients underwent salvage chemoradiation had significantly improved survival compared with chemotherapy, radiotherapy or best supportive care. For patients with locoregional recurrence, the 1-, 3-year overall survival (OS) rates were statistically higher in patients received salvage chemoradiation than radiotherapy (1-year OS, 70.0% vs. 55.2%, 3-year OS, 41.9% vs. 23.5%, p=0.045). Patients received chemotherapy had 1-year OS of 0%.

Data of 218 cases of our hospital indicated patients received radiation dose > 54Gy had a significantly longer median overall survival time of 21.2 months compared with 11.3 months in patients had <54Gy. The optimal radiation dose should be further investigated.

The recurrence pattern of patients with esophageal cancer after esophagectomy mainly consist of supraclavicular and mediastinal lymph nodes. For patients recurred after radical surgery, prophylactic irradiation to high-risk lymph node regions should be considered. The study use simultaneously integrated boost (SIB) intensity-modulated radiation therapy (IMRT) in this trial, which made different radiation dose to recurrent tumor and high-risk lymph node regions possible.

The aim of the study is to evaluate the efficacy and safety of chemoradiation therapy in patients with recurrences after radical surgery or palliative surgery. Patients were further assigned to receive elective field irradiation (ENI) or involved field irradiation (IFI) according to tumor size, tumor location and time-to-recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Locoregional recurrence after radical surgery;
* Positive resection margin (R1/R2) after surgery;
* Out-of-field recurrence after adjuvant chemoradiation or radiotherapy;
* Recurrence after adjuvant chemotherapy;
* No prior therapy after recurrence;
* Age 16-70 years;
* KPS>70;
* No history of drug allergy;
* Sufficient liver and kidney functions;
* White blood cell count > 4.0*10^9/L.

Exclusion Criteria:

* Age>70 or <16 years;
* Pregnancy or lactation;
* History of drug allergy;
* Declining informed consent;
* Insufficient liver or kidney functions, or abnormal CBC test;
* Severe cardiovascular diseases, infections, active ulcerations, diabetes mellitus with unstable blood sugar, mental disorders.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
1-, 2-, 3-year overall survival | From treatment initiation to death from any cause or censor, assessed up to 36 months
  Overall survival

SECONDARY OUTCOMES:
1-, 2-, 3-year local progression-free survival | From treatment initiation to first documented local progression or death or censor, assessed up to 36 months
  Local progression-free survival
1-, 2-, 3-year progression-free survival | From treatment initiation to first documented progression or death or censor, assessed up to 36 months
  Progression-free survival
Simultaneously integrated boost radiation therapy completion rate | During chemoradation, assessed up to 60 days
  Radiation therapy completion rate
Toxicities according to RTOG and CTCAE criteria, including hematological and non-hematological toxicities | Assessed within 3 months from initiation of chemoradiaiton (acute), and 3 months after initiation of chemoradiation (late), according to RTOG and CTCAE criteria, including hematological and non-hematological toxicities
  Toxicities of chemoradiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chang X, Deng L, Ni W, Li C, Han W, Gao LR, Wang S, Zhou Z, Chen D, Feng Q, Liang J, Bi N, Lv J, Gao S, Mao Y, Xue Q, Xiao Z. Salvage chemoradiation therapy for recurrence after radical surgery or palliative surgery in esophageal cancer patients: a prospective, multicenter clinical trial protocol. BMC Cancer. 2020 Sep 14;20(1):877. doi: 10.1186/s12885-020-07315-0. PMID 32928136